CLINICAL TRIAL: NCT06730165
Title: Comparison of the Effect of Transcutaneous Auricular Vagus and Trigeminal Nerve Stimulation on Heart Rate Variability
Brief Title: Comparison of Transcutaneous Auricular Vagus and Trigeminal Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Asst. Prof., Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: Study0009
Record Dates: First submitted 2024-11-22; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: Vagus Nerve Stimulations; Trigeminal Nerve Stimulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcutaneous Auricular Vagus Nerve Stimulation (Active Comparator): Transcutaneous vagus nerve stimulation through the tragus and concha in the ear, Frequency: 25 Hertz, Duration: 20 minutes
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Transcutaneous Auricular Trigeminal Nerve Stimulation (Active Comparator): Transcutaneous auricular trigeminal nerve stimulation, Frequency: 25 Hertz, Duration: 20 minutes
  Interventions: Device: Transcutaneous Auricular Trigeminal Nerve Stimulation
- Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham Comparator): Sham Transcutaneous Auricular Vagus Nerve Stimulation, The device is switched on but the current intensity is off, Duration: 20 minutes
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- Sham Transcutaneous Auricular Trigeminal Nerve Stimulation (Sham Comparator): Sham Transcutaneous Auricular Trigeminal Nerve Stimulation, The device is switched on but the current intensity is off, Duration: 20 minutes
  Interventions: Device: Transcutaneous Auricular Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Stimulation of the vagus nerve through the tragus and concha in the ear
  Arms: Sham Transcutaneous Auricular Vagus Nerve Stimulation; Transcutaneous Auricular Vagus Nerve Stimulation
Device: Transcutaneous Auricular Trigeminal Nerve Stimulation — Stimulation of the trigeminal nerve via the auriculotemporal nerve with a clip electrode from the upper auricle
  Arms: Sham Transcutaneous Auricular Trigeminal Nerve Stimulation; Transcutaneous Auricular Trigeminal Nerve Stimulation

SUMMARY:
The aim of this study was to compare the results between transcutaneous auricular vagus nerve stimulation and trigeminal nerve stimulation with the results obtained from heart rate variability, pulse and blood pressure measurements and to reveal which method is more effective in autonomic nervous system neuromodulation.

Hypotheses of the study:

H0: Vagus nerve stimulation is more effective than trigeminal nerve simulation in terms of heart rate variability.

H1: Trigeminal nerve stimulation is more effective than vagus nerve simulation in terms of heart rate variability.

DETAILED DESCRIPTION:
In this study, 80 healthy participants (40 males, 40 females) aged between 20-50 years were randomized (www.randomizer.org) into four groups by computer software. After randomisation, one group was received transcutaneous vagus nerve stimulation inside the ear, while the other group was received trigeminal nerve stimulation above the ear.The third group received sham transcutaneous vagus nerve stimulation and the fourth group received sham trigeminal nerve simulation. Heart rate variability, pulse rate and blood pressure measurements were performed to determine which stimulation method is more effective. Heart rate variability was analysed with Kubios HRV programme after the 5-minute short measurement method. SNS, PNS and Stress Index and LF, HF and LF/HF parameters were evaluated in heart rate variability sub-parameters.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years of age or older,
* Not having any acute or chronic disease.

Exclusion Criteria:

* Having any acute or chronic disease,
* Having previously undergone vagus nerve stimulation or trigeminal nerve stimulation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Pre-intervention and immediately after the intervention
  5 minutes of heart rate variability was measured.

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | Pre-intervention and immediately after the intervention
  Systolic and diastolic blood pressure was measured with an electronic blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Ozoran, Prof., Study Chair — Dean of the Health Sciences Faculty
Locations (1):
- Avrasya University, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Li SY, Wang D, Wu MZ, He JK, Zhang JL, Zhao B, Hou LW, Wang JY, Wang L, Wang YF, Zhang Y, Zhang ZX, Rong PJ. Transcutaneous Auricular Vagus Nerve Stimulation: From Concept to Application. Neurosci Bull. 2021 Jun;37(6):853-862. doi: 10.1007/s12264-020-00619-y. Epub 2020 Dec 23. PMID 33355897
- [Background] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Background] Milby AH, Halpern CH, Baltuch GH. Vagus nerve stimulation for epilepsy and depression. Neurotherapeutics. 2008 Jan;5(1):75-85. doi: 10.1016/j.nurt.2007.10.071. PMID 18164486
- [Derived] Percin A, Ozden AV, Yenisehir S, Albayrak HE. Autonomic Effects of Transcutaneous Auricular Vagus and Trigeminal Nerve Stimulation: A Randomized, Sham-Controlled, and Single-Blind Study. Neuromodulation. 2025 Oct 27:S1094-7159(25)01038-4. doi: 10.1016/j.neurom.2025.09.312. Online ahead of print. PMID 41143755